CLINICAL TRIAL: NCT06051838
Title: Prognostic Value of Tumor Deposits for Patients With Papillary Thyroid Carcinoma: a Retrospective Cohort Study
Brief Title: Prognostic Value of Tumor Deposits for Patients With Papillary Thyroid Carcinoma
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-326
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Exploring the Prognostic Value of Tumor Deposits PTC Patients
Keywords: tumor deposits, extranodal extension, papillary thyroid carcinoma, lymph node metastasis, prognosis.
MeSH Terms: conditions — Extranodal Extension; Thyroid Cancer, Papillary; Lymphatic Metastasis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TD cohort: Tumor deposits (TD) positive group, which was determinded by the pathologists at department of pathology. Any tumor mass, either circumscribed or with irregular contours, devoid of lymph node architecture was identified as a tumor deposit.
  Interventions: Procedure: surgery
- Non-TD cohort: Tumor deposits (TD) negative group, which was determinded by the pathologists at department of pathology. No visiblet umor mass, either circumscribed or with irregular contours, devoid of lymph node architecture in the sections of specimens from these patients.
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — if the patients is TD positive, we recommond careful surgery and pathological examination.

SUMMARY:
Tumor deposits (TD), nodules in the peritumoral adipose tissue with no architectural residue of lymph node, which is a definition often being confusing to the extranodal extension (ENE), have been described in several malignancies and linked to a worse prognosis. In gastric cancer and colon cancer, TD and ENE should be distinguished and collected separately in 8th AJCC manual. However, in thyroid cancer, TD as a collection variable was absence in both the 8th AJCC manual and the 2015 ATA guideline. This is a study that revealed the presence of TD by reviewing a large number of papillary thyroid carcinoma (PTC) specimens and explored its prognostic value by constructing a nomogram to accurately predict disease-free survival in PTC patients.

ELIGIBILITY:
Inclusion Criteria:

(1) patients with histopathologically confirmed PTC and sections stored in the pathology department; (2) patients underwent lobectomy or total thyroidectomy and central lymph node dissection with or without lateral neck dissection; (3) patients cooperated to provide follow-up information after surgery.

Exclusion Criteria:

(1) patients with previous history of neck irradiation or other systematic cancers; (2) patients died of unrelated diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Five hundred and forty-one PTC patients were enrolled in this study. Their clinicopathological characteristics are shown in Table 1. The study population consisted of 186 (34.4%) males and 355 (65.6%) females, with median (IQR) age of 40 [31 to 50]. Of the patients, 13.3% were older than 55 years old. Median follow-up time after surgery was 35 months (IQR, 27 to 42 months).
  TD was identified in 87 (16.1%) patients (TD-positive cohort). The rest of patients (n = 454, 83.9%) were not found with TD (Non-TD cohort). Female proportion was smaller in the TD positive cohort than in Non-TD cohort (51.7% vs 68.3%; p = 0.009). TD cohort has a higher proportion of age over 55 years than Non-TD cohort (20.7% vs 11.9%, p = 0.041). No differences in body mass index (BMI) (23.03 vs 23.22 kg/m2, p = 0.221) was observed between the TD cohort and Non-TD cohort.
Sampling Method: Non-Probability Sample
Enrollment: 541 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
disease-free survival (DFS) after diagnosis | between 2015 and 2021
  The primary outcome was disease-free survival (DFS) after diagnosis, with endpoints as tumor locoregional recurrence, distant metastasis, and disease-specific death. If a patient was deceased, the cause of death was confirmed by the death certificate or the hospitalization record to identify disease-specific death.

SECONDARY OUTCOMES:
Disease recurrence | between 2015 and 2021
  Disease recurrence was defined as recurrent or persistent PTC identified with standard biochemical, cytological, histological, and radiographical criteria. In this study, tumor locoregional recurrence was defined as combined biochemical (serum thyroglobulin) and structural recurrences.

CONTACTS AND LOCATIONS:
Overall Officials: Shangtong Lei, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided